CLINICAL TRIAL: NCT00178503
Title: ADHD Symptoms in Autism: Cognition, Behavior, Treatment
Brief Title: Methylphenidate for Attention Deficit Hyperactivity Disorder and Autism in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deborah Pearson, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH072263 (NIH); R01MH072263 (NIH); DDTR B2-NDA
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Autism; Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MPH Trial-Placebo (Placebo Comparator): 24 Participants with ASD-ADHD underwent 1 week of placebo in the MPH treatment phase
  Interventions: Other: Placebo
- MPH Trial: Low Dose (Active Comparator): 24 Participants with ASD-ADHD underwent 1 week at a low dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
  Interventions: Drug: Methylphenidate-extended release; Drug: Methylphenidate-immediate release
- MPH Trial: Med Dose (Active Comparator): 24 Participants with ASD-ADHD underwent 1 week at a medium dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
  Interventions: Drug: Methylphenidate-extended release; Drug: Methylphenidate-immediate release
- MPH Trial: High Dose (Active Comparator): 24 Participants with ASD-ADHD underwent 1 week at a high dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
  Interventions: Drug: Methylphenidate-extended release; Drug: Methylphenidate-immediate release

INTERVENTIONS:
Drug: Methylphenidate-extended release — Methylphenidate-extended release was taken in the morning of the MPH treatment trial. Each participant underwent 1 week of the each of the doses as determined by body weight. The lower body weight group (20 to 24 kg/44 to 52.8 lbs) took 10 mg Ritalin LA to 20 mg. The medium body weight group (25 to 33 kg/55 to 72.6 lbs) took from 10 mg Ritalin LA to 30 mg. The higher body weight group (34 to 59 kg/74.8 to 129.8 lbs) took 20 mg Ritalin LA to 40 mg.
  Other Names: Ritalin LA
  Arms: MPH Trial: High Dose; MPH Trial: Low Dose; MPH Trial: Med Dose
Drug: Methylphenidate-immediate release — Methylphenidate-immediate release was taken in the late afternoon. Each participant underwent 1 week at each of the 3 dose levels as determined by body weight. The lower body weight group (20 to 24 kg/44 to 52.8 lbs) took 2.5 mg IR-MPH and 2 weeks of 5 mg. The medium body weight group (25 to 33 kg/55 to 72.6 lbs) took 2 weeks of 5 mg IR-MPH and 1 week of 10 mg. The higher body weight group (34 to 59 kg/74.8 to 129.8 lbs) took 1 week of 5 mg IR-MPH and 2 weeks of 10 mg.
  Arms: MPH Trial: High Dose; MPH Trial: Low Dose; MPH Trial: Med Dose
Other: Placebo — Participants will take a placebo for 1 full week of the randomized drug trial. They will take one capsule in the morning and one capsule in the afternoon.
  Arms: MPH Trial-Placebo

SUMMARY:
This study examined the cognitive and behavioral differences in children who have an autism spectrum disorder (ASD) with or without additional symptoms of ADHD. The study also examined the effectiveness of a range of doses of methylphenidate in improving cognitive and behavioral outcomes in children with both ASD and ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is a major comorbid psychiatric disorder in children with Autism Spectrum Disorders (ASD) that significantly undermines behavioral, social, and emotional adjustment. Although the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) does not specifically allow for a comorbid diagnosis of ADHD with ASD, many children with an ASD manifest symptoms of ADHD and are treated for it with stimulants or other medication. The few studies on ADHD in ASD have not consistently established its cognitive and behavioral manifestations, or the optimal parameters for treatment. The proposed project will address these issues through studies of cognitive and behavioral functioning in children with ASD, with and without ADHD, and through a study of medication treatment of ADHD symptoms in autism.

Participants between the ages of 7 to 12 with an autism spectrum disorder participated in the initial phase of the study to examine the nature and effects of ADHD symptoms on behavioral and cognitive functioning. Participants underwent an initial psychological testing session that included standardized measures of intellectual, adaptive behavior, language, behavioral, and emotional functioning, along with standardized diagnostic measures to confirm their diagnoses of ASD and/or ADHD (Visit 1). Children with intelligence quotients (IQs) below 50 or greater than 130 or with major sensory, motor, neurological, genetic, or psychiatric disorders that may interfere with testing were be excluded. The participants who meet eligibility criteria completed computerized tasks of attentional functioning in a second visit (Visit 2).

A subset of the children meeting criteria for the ASD/ADHD group (N=24) participated in a six-week randomized double-blind, placebo-controlled treatment trial using various doses (low, medium, or high dose) of methylphenidate (MPH). Children participated in the treatment trial will be those who qualified based on the initial phase and who do not have any physical contraindications to MPH (e.g., history of MPH intolerance). In each week of the treatment trial, the children took one of the three doses of MPH or a placebo. At the end of each week the child were evaluated in the clinic by including a medical check-up, parent interviews about the child's behavior and functioning that week, and computerized cognitive testing. Additionally, the child's parent and teacher completed questionnaires about the child's behavior each week, so that the child's home and school behaviors at each MPH dose could be assessed.

ELIGIBILITY:
Inclusion Criteria:

Autism/ADHD Group:

* DSM-IV diagnosis of autistic disorder, as per the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS)
* Child manifests current symptoms of ADHD

Autism/non-ADHD Group:

* Meets the diagnostic criteria for autism, as above, but does not meet the diagnostic criteria for ADHD

Exclusion Criteria:

In both groups, exclusion criteria will include:

* Sensory or motor deficits sufficient to interfere with testing (e.g., blindness, severe cerebral palsy)
* Serious neurological disorders (e.g., epilepsy, stroke)
* Down syndrome, fragile X syndrome, Tourette syndrome, or fetal alcohol syndrome
* Bipolar disorder or a family history of bipolar disorder in a first-degree relative
* Other serious psychopathology that resulted in psychiatric hospitalization (e.g., for psychotic episode). The investigators will screen for this using the Diagnostic Interview for Children and Adolescents (DICA)-IV, and getting a complete developmental/medical history
* Serious physical handicaps that would interfere with performance on laboratory tasks
* IQ less than 50 and greater than 130
* Verbal mental age (VMA) less than 36 months (to exclude participants unable to understand simple task instructions)

In the autism/ADHD group, further exclusion criteria apply to the MPH trial:

* History of intolerance to MPH
* Weight less than 20 kg or greater than 59 kg (less than 44 pounds or greater than 130 pounds)
* Concomitant use of dextroamphetamine preparations (Dexedrine, Dextrostat), mixed amphetamine salts (Adderall XR), other MPH preparations (e.g., Concerta, Metadate); venlafaxine, bupropion, atomoxetine, guanfacine, modafinil.
* Concomitant use of any herbal preparations
* Medical condition for which stimulants are contraindicated (e.g., high blood pressure)
* Past treatment failure on a methylphenidate trial

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Pearson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January of 2006 to March of 2010. Sources of recruitment included our UT Department of Psychiatry Clinics, research registry, along with community referrals from local agencies, parent groups, and schools.
Pre-assignment Details: 129 children completed the initial psychological/screening assessment to confirm study eligibility. Of those 129 children, 94 children met full inclusion/exclusion criteria for the initial phase project. Of these, 28 were invited to participate in the MPH trial and 24 of these children were randomized into the trial.
Groups:
- MPH Trial: 24 participants with autism spectrum disorder and ADHD underwent a randomized, placebo-controlled, cross-over designed trial, which included: 1 week of placebo, 1 week of low dose methylphenidate, 1 week of medium dose methylphenidate, 1 week of high dose methylphenidate.
Period: MPH Trial: Placebo
Arm/Group | MPH Trial
Started | 24
Completed | 24
Not Completed | 0
Period: MPH Trial: Low Dose
Arm/Group | MPH Trial
Started | 24
Completed | 24
Not Completed | 0
Period: MPH Trial: Med Dose
Arm/Group | MPH Trial
Started | 24
Completed | 24
Not Completed | 0
Period: MPH Trial: High Dose
Arm/Group | MPH Trial
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MPH Trial: 24 Participants with ASD-ADHD underwent 1 week of placebo, 1 week of Low dose, 1 week of Medium dose, and 1 week of High dose in the MPH treatment phase
Arm/Group | MPH Trial
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Conners' Teacher ADHD Index T Score by Dose
Description: The ADHD Index of the Conners' Teacher Rating Scale-Revised (CTRS-R) assesses symptoms associated with ADHD, including inattentiveness, hyperactivity and impulsivity. Lower T-scores on this subscale are associated with milder ADHD symptoms. T-scores have a mean of 50 and a SD of 10. Thus, T-scores of 70+ (i.e., 2 SD's over the mean) on the ADHD Index are suggestive of very significant ADHD symptomatology. Treatment-related changes of 5+ points are considered to be significant.
Time Frame: Measured at each dosing week of the drug trial (placebo, low, medium, high)
Population: Although there were 24 participants who completed the trial, teacher ratings were only available for 18 participants due to 6 children being seen during the summer months.
Measure: Mean (Standard Deviation); unit: Units on a scale (T-scores)
Groups:
- MPH Trial-Placebo Week: All 24 participants with ASD-ADHD underwent 1 week of placebo in the MPH treatment phase
- MPH Trial: Low Dose Week: All 24 participants with ASD-ADHD underwent 1 week at a low dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: Med Dose Week: All 24 participants with ASD-ADHD underwent 1 week at a medium dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: High Dose Week: All 24 participants with ASD-ADHD underwent 1 week at a high dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phasephase
Arm/Group | MPH Trial-Placebo Week | MPH Trial: Low Dose Week | MPH Trial: Med Dose Week | MPH Trial: High Dose Week
Number analyzed (Participants) | 18 | 18 | 18 | 18
Units on a scale (T-scores) | 72.8 (12.0) | 63.1 (11.2) | 63.6 (10.4) | 61.5 (13.0)
Statistical Analysis 1: Comparison: MPH Trial-Placebo Week vs MPH Trial: Low Dose Week vs MPH Trial: Med Dose Week; Data were analyzed using SPSS-PC repeated measures one-way analysis of variance (ANOVA), with MPH dosing regimen as the within-subjects variable; Test type: Superiority or Other; p = .001, ANOVA; Linear trend P value = .000

2. Primary Outcome: Mean Continuous Performance Test (CPT)-Commission Errors by Dose
Description: CPT is a measure of sustained attention using nonverbal stimuli (pictures). Participants are asked to click on the witch (target), which appears for 25% of the trials. Commission errors are measured by number of times they click for the non-target items.
Time Frame: Measured at each dosing week of the drug trial (placebo, low, medium, high)
Measure: Mean (Standard Deviation); unit: Total Errors
Groups:
- MPH Trial-Placebo Week: Participants with ASD-ADHD underwent 1 week of placebo in the MPH treatment phase
- MPH Trial: Low Dose Week: Participants with ASD-ADHD underwent 1 week at a low dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: Med Dose Week: Participants with ASD-ADHD underwent 1 week at a medium dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: High Dose Week: Participants with ASD-ADHD underwent 1 week at a high dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
Arm/Group | MPH Trial-Placebo Week | MPH Trial: Low Dose Week | MPH Trial: Med Dose Week | MPH Trial: High Dose Week
Number analyzed (Participants) | 24 | 24 | 24 | 24
Total Errors | 2.75 (3.49) | 1.11 (1.91) | 1.18 (1.71) | 1.24 (2.27)
Statistical Analysis 1: Comparison: MPH Trial-Placebo Week vs MPH Trial: Low Dose Week vs MPH Trial: Med Dose Week vs MPH Trial: High Dose Week; Test type: Superiority or Other; p = .005, ANOVA; Linear p = .005

3. Secondary Outcome: Mean Conners' Parent ADHD Index T Score by Week
Description: The ADHD Index of the Conners' Parent Rating Scale-Revised (CPRS-R) assesses symptoms associated with ADHD, including inattentiveness, hyperactivity and impulsivity. Lower T-scores on this subscale are associated with milder ADHD symptoms. T-scores have a mean of 50 and a SD of 10. Thus, T-scores of 70+ (i.e., 2 SD's over the mean) on the ADHD Index are suggestive of very significant ADHD symptomatology. Treatment-related changes of 5+ points are considered to be significant.
Time Frame: Measured at each dosing week of the drug trial (placebo, low, medium, high)
Measure: Mean (Standard Deviation); unit: Units on a scale (T-scores)
Groups:
- MPH Trial: Low Dose Week: Participants with ASD-ADHD who will undergo 1 week at a low dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
Arm/Group | MPH Trial-Placebo Week | MPH Trial: Low Dose Week | MPH Trial: Med Dose Week | MPH Trial: High Dose Week
Number analyzed (Participants) | 24 | 24 | 24 | 24
Units on a scale (T-scores) | 70.1 (12.0) | 64.9 (9.3) | 62.3 (10.0) | 59.9 (10.5)
Statistical Analysis 1: Comparison: MPH Trial-Placebo Week vs MPH Trial: Low Dose Week vs MPH Trial: Med Dose Week vs MPH Trial: High Dose Week; Test type: Superiority or Other; p < .001, ANOVA; Linear p = .000

ADVERSE EVENTS:
Time Frame: over 4 weeks of the trial
Groups:
- MPH Trial-Placebo: Participants with ASD-ADHD who will undergo 1 week of placebo in the MPH treatment phase
- MPH Trial: Low Dose: Participants with ASD-ADHD who will undergo 1 week at a low dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: Med Dose: Participants with ASD-ADHD who will undergo 1 week at a medium dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
- MPH Trial: High Dose: Participants with ASD-ADHD who will undergo 1 week at a high dose of Methylphenidate-extended release and Methylphenidate-immediate release in the MPH treatment phase
Arm/Group | MPH Trial-Placebo | MPH Trial: Low Dose | MPH Trial: Med Dose | MPH Trial: High Dose
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 13/24 | 15/24 | 17/24 | 15/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MPH Trial-Placebo (N=24) | MPH Trial: Low Dose (N=24) | MPH Trial: Med Dose (N=24) | MPH Trial: High Dose (N=24)
Repetitive Behaviors (Psychiatric disorders) | 12 | 11 | 12 | 9
Repetitive Language (Psychiatric disorders) | 12 | 9 | 12 | 9
Irritability (Psychiatric disorders) | 11 | 8 | 8 | 7
Anxiety (Psychiatric disorders) | 4 | 4 | 6 | 2
Sadness (Psychiatric disorders) | 3 | 2 | 4 | 1
Euphoria (Psychiatric disorders) | 1 | 0 | 0 | 0
Hair or skin pulling (Psychiatric disorders) | 2 | 1 | 1 | 2
Facial or body tics (Psychiatric disorders) | 0 | 1 | 1 | 2
Unusual Blinking (Psychiatric disorders) | 0 | 1 | 1 | 0
Trouble sleeping (Psychiatric disorders) | 5 | 7 | 12 | 9
skin rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Stomach ache (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Loss of Appetite (Gastrointestinal disorders) | 1 | 7 | 9 | 9
Dry Mouth (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Staring (Nervous system disorders) | 4 | 0 | 2 | 1
Racing heart (Cardiac disorders) | 0 | 0 | 1 | 0
Drowsiness (Nervous system disorders) | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 4 | 2
Fever (Immune system disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
We did not have teacher behavioral data for all of the children because some of them were seen during the summer, when teacher input was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No